CLINICAL TRIAL: NCT05330442
Title: Delivering Written Exposure Therapy for PTSD in Underserved Primary Care Settings
Brief Title: Building Experience for Treating Trauma and Enhancing Resilience (BETTER)
Acronym: BETTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Boston University (Other); Clinical Directors Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH123585
Record Dates: First submitted 2022-04-01; First posted 2022-04-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: PTSD; brief psychotherapy; collaborative care; Federally Qualified Health Centers (FQHCs); primary care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Matched pairs of health centers/FQHCs will be randomized to either CoCM alone or to CoCM+WET.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not know which are patients within health centers are assigned to because they will be independent of the participant recruitment coordinators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoCM alone (No Intervention): In the CoCM alone arm, participants will have access to treatment as usual from the CM.
- CoCM+WET (Experimental): In the CoCM+WET intervention arm, patients will be encouraged to receive WET.
  Interventions: Behavioral: Written Exposure Therapy (WET)

INTERVENTIONS:
Behavioral: Written Exposure Therapy (WET) — The WET protocol for primary care settings consists of six, 30-minute sessions. The first session consists of psychoeducation of PTSD and treatment rationale. Written narratives are conducted in sessions 2-6, following specific writing instructions and 20 minutes of writing in each session.
  Arms: CoCM+WET

SUMMARY:
Posttraumatic stress disorder (PTSD) is a significant problem among underserved populations who receive care in community health centers. Several evidence-based psychotherapies for PTSD are not practical given the time and resources required for these approaches. This research will examine whether Written Exposure Therapy (WET), a brief and well-tolerated therapy approach, delivered within collaborative primary care is effective and can be implemented successfully within a collaborative care (CC) intervention. The primary aims of the proposed study are to evaluate the effectiveness and implementation of delivering WET into CoCM to improve the management of PTSD among underserved primary care patients in Federally Qualified Health Centers (FQHCs).

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) results in substantial costs to society is highly prevalent among adults. Importantly, the prevalence PTSD within primary care settings is even higher than the general population as primary care is the setting to which individuals with PTSD most often present. Evidence-based psychotherapies (EBPs) for PTSD are available but dissemination within real world settings is fraught with challenges because these therapies require 10-15, lengthy treatment sessions and extensive therapist training to implement, and these treatments are not feasible within primary care settings given the limited time resources. Consequently, there are multiple barriers to accessing EBPs for PTSD. Efforts to integrate mental health services within primary care for PTSD though collaborative care management (CoCM) interventions are rapidly expanding and have been shown to be effective in the treatment of depression and anxiety. However, the evidence for PTSD is limited due to the time intensive nature of the PTSD therapy approaches that have been examined. An efficient PTSD treatment approach is needed to address the treatment needs of individuals with PTSD presenting to primary care. Written exposure therapy (WET) is a brief EBP that provides an alternative to more intensive EBPs. Recent studies of WET have yielded positive outcomes and have shown it to be non-inferior when directly compared to more time intensive PTSD EBPs, but WET has not yet been examined within the primary care environment. The primary aims of the proposed study are to evaluate the effectiveness and implementation of delivering WET into CoCM to improve the management of PTSD among underserved primary care patients in Federally Qualified Health Centers (FQHCs). The pragmatic cluster-randomized study will use a hybrid effectiveness-implementation design. Twelve FQHCs will be randomized to either CoCM plus WET (CoCM+WET) or CoCM alone and 60 patients within each FQHC will be screened for eligibility. The investigators will use the RE-AIM framework (for Reach, Efficacy/Effectiveness, Adoption, Implementation, & Maintenance) to evaluate the effectiveness and implementation process of the CoCM+WET intervention using mixed methods. To examine effectiveness and potential mediators and moderators of the intervention, the investigators will administer assessments at baseline, 3- and 12-month follow-up. To assess implementation, the investigators will use clinic process data and clinic staff interviews pre- and post-intervention. This study has the potential to substantially impact practice and public health by validating the effectiveness and feasibility of delivering a brief trauma-focused EBP embedded within CoCM in primary care to improve PTSD outcomes for underserved patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are 18 years of age or older, speak English or Spanish, have a scheduled or walk-in appointment with a participating primary care provider (PCP), have no obvious physical or cognitive impairment that would make them unable to complete the assessment (as indicated by confusion or inability to understand the questions), and consider the FQHC to be their usual source of care.

Exclusion Criteria:

* Patients will be excluded if they have active psychosis (as indicated by inability to concentrate, having delusions or hallucinations) or high suicide risk (as indicated by having a current plan or means).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist, version 5 (PCL-5) | baseline
  PTSD symptoms (total score) and provisional diagnosis anchored to the worst traumatic event
PTSD Checklist, version 5 (PCL-5) | 3-months
  PTSD symptoms (total score) and provisional diagnosis anchored to the worst traumatic event
PTSD Checklist, version 5 (PCL-5) | 12-months
  PTSD symptoms (total score) and provisional diagnosis anchored to the worst traumatic event

SECONDARY OUTCOMES:
Patient Health Questionnaire, 8 items (PHQ-8) | baseline
  Depression symptoms (total score) and probable diagnosis
Patient Health Questionnaire, 8 items (PHQ-8) | 3-months
  Depression symptoms (total score) and probable diagnosis
Patient Health Questionnaire, 8 items (PHQ-8) | 12-months
  Depression symptoms (total score) and probable diagnosis
Veterans RAND 12-item Health Survey (VR-12) | baseline
  Mental and physical health functioning component scores
Veterans RAND 12-item Health Survey (VR-12) | 3-months
  Mental and physical health functioning component scores
Veterans RAND 12-item Health Survey (VR-12) | 12-months
  Mental and physical health functioning component scores

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Higby, Study Director — RAND
Locations (10):
- United States (10):
  - Oak Orchard Health Center (Albion), Albion, New York
  - Brownsville Health Center (Genesis and Ashford - BGA), Brooklyn, New York
  - Brownsville Health Center (Main), Brooklyn, New York
  - Bedford Stuyvesant Family Health Center (Main), Brooklyn, New York
  - Bedford Stuyvesant Family Health Center (Sterling and Broadway), Brooklyn, New York
  - Oak Orchard Health (Pembroke), Corfu, New York
  - Open Door Family Medical Center (Brewster/Ossining), Ossining, New York
  - Open Door Family Medical Center (Mamaroneck//Port Chester), Port Chester, New York
  - OIC Family Medical Center (Fairview), Rocky Mount, North Carolina
  - OIC Family Medical Center (Happy Hill), Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the research programmer will upload participant data to the NIMH Data Archive.
Supporting Information: Study Protocol, ICF
Time Frame: May 2026
Access Criteria: Data will be shared through the NIMH Data Archive

REFERENCES:
- [Background] Meredith LS, Wong EC, Marx BP, Han B, Korn AR, Tobin JN, Cassells A, Williamson S, Franco M, Overa CC, Holder T, Lin TJ, Sloan DM. Design of a hybrid implementation effectiveness cluster randomized controlled trial of delivering written exposure therapy for PTSD in underserved primary care settings. Contemp Clin Trials. 2024 Mar;138:107435. doi: 10.1016/j.cct.2024.107435. Epub 2024 Jan 9. PMID 38211725

DOCUMENTS (1):
  • Informed Consent Form (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05330442/ICF_000.pdf